CLINICAL TRIAL: NCT06185257
Title: Electroencephalographic Changes in Nonconvulsive Children With Chronic Renal Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khloud Abd-elnasser Saleh Seif, Principal invistigator, Assiut University
Other Study IDs: Electroencephalographic change
Record Dates: First submitted 2023-11-20; First posted 2023-12-29 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Chronic Renal Disease and Nephrotic Syndrome
MeSH Terms: conditions — Renal Insufficiency, Chronic; Nephrotic Syndrome | interventions — Electroencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient with chronic kidney disease under dialysis
  Interventions: Device: EEG
- Patients with nephrotic syndrome
  Interventions: Device: EEG
- C. Normal control group
  Interventions: Device: EEG

INTERVENTIONS:
Device: EEG — Methodology Subjects selected are divided into 3 groups A. Patient with chronic kidney disease under dialysis B. Patients with nephrotic syndrome
  * Patients in remission
  * Patients relapse C. Normal control group
  Detailed history including age, sex , residence ,complain, renal symptoms will be taken.
  Detailed examination, lab investigations, and treatment will be recorded
  Imaging ( EEG) , results of the three groups will be assessed and compared and lab investigation ( lipid profile of all patients) will be measured

SUMMARY:
Chronic kidney disease (CKD) arises from many heterogeneous disease pathways that alter the function and structure of the kidney irreversibly, over months or years. The diagnosis of CKD rests on establishing a chronic reduction in kidney function and structural kidney damage. The best available indicator of overall kidney function is glomerular filtration rate (GFR), which equals the total amount of fluid filtered through all of the functioning nephrons per unit of time

The definition and classification of CKD have evolved over time, but current international guidelines define CKD as decreased kidney function shown by GFR of less than 60 mL/min per 1·73 m2, or markers of kidney damage, or both, of at least 3 months duration, regardless of underlying cause . When GFR is less than 15 mL/min per 1·73m2 , a person has reached end stage kidney disease (ESKD), at which point kidney function is no longer able to sustain life over the long term. Options for patients with ESKD are kidney replacement therapy (in the form of dialysis or kidney transplantation), or conservative care (also called palliation or non-dialytic care

Encephalopathy detected in patients with chronic kidney disease results from their exposure to several factors, such as uremia, hypertension, and fluid, and electrolyte disturbances (Brouns R, DyDeyn pp,2004)

Uremic encephalopathy features include alterations of mental status (alertness and awareness alterations, poor concentration, psychosis, and hallucinations, without treatment of which stupor, and coma may develop) and motor system abnormalities, such as clouding of the sensorium as an early feature and delirium, seizures, and coma as late features (Palmer sc ,etal,2010)EEG is useful in assessing patients in uremic encephalopathy and in monitoring their progress. Electroencephalographic (EEG) findings correlate with clinical symptoms and, therefore, may be of diagnostic value. In addition, it can be useful to exclude other causes of confusion such as infection or structural abnormalities (Dijck Annemie Van,etal,2012).

The EEG in uremic encephalopathy is generally abnormal, showing generalized slowing that becomes more severe as the condition worsens. EEG in CKD usually shows irregular low voltage with slowing of the posterior dominant alpha rhythm and occasional theta bursts. Prolonged bursts of bilateral, synchronous slow and sharp waves or spike and waves are characteristic. These changes stabilize with dialysis. EEG abnormalities in uremic encephalopathy is reflected through appearance of theta waves, disappearance of normal basic rhythms and diminished reactivity of EEG to afferent stimulation and domination by generalized delta activity. All these changes are mostly appreciated in the frontal leads (Al Arieff,Philadelphia,Ssaunders,2004)(Cl fraser, Arieff,Philadelphia,2001)

A lot of studies have been done about uremic encephalopathy in acute renal failure patients. Very few data are available regarding EEG changes in CKD. This study evaluates the EEG findings in different stages of CKD.

DETAILED DESCRIPTION:
Aim of the study Evaluate electroencephalographic changes in children with chronic renal disease and nephrotic syndrome

Patient and Method include :

Methodology Subjects selected are divided into 3 groups A. Patient with chronic kidney disease under dialysis B. Patients with nephrotic syndrome

* Patients in remission
* Patients relapse C. Normal control group

Detailed history including age, sex , residence ,complain, renal symptoms will be taken.

Detailed examination, lab investigations, and treatment will be recorded

Imaging ( EEG) , results of the three groups will be assessed and compared and lab investigation ( lipid profile of all patients) will be measured

TYPE OF THE STUDY

Observational study

Sitting of the study

Assiut University children hospital Inclusion criteria

All children with chronic kidney disease and nephrotic syndrome

Exclusion criteria

* Newborn
* Patients with genetic disease Neurological disorder

Sample size Based on determining the main outcome variable, the estimated minimal required sample size is 102 patient (34 patient in each group).the sample was calculated using Gpower software 3.1.9.2.,based on the following assumptions: main outcome variable is the deference in the main value of relative power of delta band of patients with chronic kidney disease ,patients with nephrotic syndrome, and normal control group. based on clinical experience we expected to find large effect size difference between the 3 groups .main statistical test is independent t-test to detect the difference between the 3 groups Alpha=.05 Power=.95 Effect size=1.1

Statistical analysis

All statistical analysis will be performed by SPSS version 20. Mean and standard deviation will be used for descriptive statistics . for quantitative data

Ethical considerations:

1. risk-benefit ratio The EEG has been used for many years and is considered a safe procedure. The test causes no discomfort. The electrodes record activity. They do not produce any sensation. In addition, there is no risk of getting an electric shock.
2. confidenity Any data taken from the patient either from history the examination or the investigations will be very confidential
3. researsh statement Every patient subjected to this study will be informed about the procedure of the research
4. informed consent The aim of our investigation will be explained to all parents and informed written consent was taken as well • Other ethical concerns The research will be conducted only by scientifically qualified and trained personnel

ELIGIBILITY:
Inclusion Criteria:

* All children with chronic kidney disease and nephrotic syndrome

Exclusion Criteria:

* Newborn
* Patients with genetic disease Neurological disorder

Ages: 6 Months to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Electroencephalographic changes in nonconvulsive children with chronic renal disease
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-09-15 (Estimated); Primary Completion 2025-01-15 (Estimated); Study Completion 2025-01-15 (Estimated)

PRIMARY OUTCOMES:
Electroencephalographic changes in non convulsive children with chronic renal disease | one year
  Evaluate electroencephalographic changes in children with chronic renal disease and Under dialysis and without dialysis changes in wave form , amplitude of waves , symmetry,sharp waves present or not in EEG compared to normal children Under dialysis and without dialysis as wave changes in EEG compared to normal children